CLINICAL TRIAL: NCT01876147
Title: A Randomised Crossover Study to Assess the Usability of Two New Vision Tests in Patients With Low Vision, and Relationship of the Measures to Daily Living Tasks.
Brief Title: Visual and Functional Assessment in Low Vision Patients
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OxfordVA2013
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2018-10

CONDITIONS: Retinitis Pigmentosa; Age-related Macular Degeneration; Optic Nerve Pathology; Inherited Retinal Dystrophies
Keywords: Low vision; Vision testing; Retinitis Pigmentosa; AMD; Visual acuity; Poor vision; Quantification
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Vision, Low; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Order of vision tests 1: Undergo testing with BRVT first, FrACT second.
- Order of vision tests 2: Undergo testing with FrACT first, BRVT second.

SUMMARY:
Vision testing is a fundamental part of every optometry and ophthalmology assessment. Traditional vision testing charts are not able to measure vision below a certain level. Vision in this range is classified as counting fingers (CF), hand movements (HM) and light perception (LP). These measures are not very accurate or easily quantifiable. They are also poorly understood in terms of impact on quality of life. This study aims to assess new methods for measuring the vision of patients with very low vision.

DETAILED DESCRIPTION:
Assessing very low vision accurately is becoming increasingly important with the increase in research in this area, such as using retinal implants to restore vision. Without being able to accurately measure the change in vision before and after treatment, it is not possible to fully assess the effect of treatment.

The Freiburg Vision Test (FrACT) is a computer based test developed to assess patients down to the LP level. It has been used in research in recent years. The FrACT is suitable for research but is not suitable for a clinical setting. The Berkeley Rudimentary Vision Test (BRVT) works on a similar principal as the FrACT but consists of hand held cards shown to the patient. Little work has been completed on how well the BRVT test works. Results from FrACT and BRVT will be compared in a group of patients with very low vision. This is important to establish how easily research results can be applied to a clinical setting.

Patients will also be asked to complete a daily living survey to better understand the impact of such poor vision on the ability to carry out day to day tasks. This understanding will help guide low vision services for patients as well as help direct low vision research to achieve a useful level of functional vision.

ELIGIBILITY:
Inclusion Criteria:

* Snellen VA or equivalent ≤ 6/60 in both eyes
* Patient has capacity to give consent and to undertake vision tests

Exclusion Criteria:

* Diagnosis of functional vision loss
* Unwilling and/or unable to sign informed consent and complete the vision tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low vision attending outpatient clinics in Oxford Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of VA measured with FrACT and BRVT vision tests | Single visit

SECONDARY OUTCOMES:
Relationship between VA and ability to carry out daily living tasks. | Single time point
  Results from a daily living skills survey will be related to VA measured by FrACT testing.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] Jolly JK, Gray JM, Salvetti AP, Han RC, MacLaren RE. A Randomized Crossover Study to Assess the Usability of Two New Vision Tests in Patients with Low Vision. Optom Vis Sci. 2019 Jun;96(6):443-452. doi: 10.1097/OPX.0000000000001380. PMID 31058709
- See also: Related Info — https://www.ndcn.ox.ac.uk/divisions/nlo/